CLINICAL TRIAL: NCT05289505
Title: Prospective and Monocentric Pilot Study of the Evaluation of the Music Delivered by the Music-Care Device on the Level of Anxiety Felt During External Radiotherapy Sessions
Brief Title: Evaluation of Music on the Level of Anxiety Felt During External Radiotherapy Sessions
Acronym: MUSIC-RT
Status: Completed | Type: Observational
Sponsor: Center Eugene Marquis (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-6-63-004; 2021-A00597-37 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2022-01-25; First posted 2022-03-21 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2022-09

CONDITIONS: Radiotherapy Side Effect
Keywords: Anxiety
MeSH Terms: conditions — Radiation Injuries; Anxiety Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective phase: This prospective phase involves all patients with an initial HADS score > 7 and initiating treatment in the radiotherapy department. The treatment sessions will be performed with music, using the MUSIC-CARE device. In the event of technical problems, unavailability of equipment, or the patient's wishes, some radiotherapy sessions may be conducted without music. Nevertheless, a minimum of one weekly session with music is required for the analysis of the study.
  Interventions: Device: MUSIC-CARE

INTERVENTIONS:
Device: MUSIC-CARE — This device allows the listening of music using different sequences of instrumental music created specifically, and using principles based on hypno-analgesia, that is to say the association of hypnotic techniques and approaches to help or analgesic, medicated or not. It consists of a tablet application containing instrumental music pieces, specially created and recorded for Music-Care. Each piece is at least 20 minutes long. The music can be played through headphones or speakers.

SUMMARY:
This is a prospective study with a historical comparator. Each of the prospective study endpoints will be compared to data collected retrospectively in patients treated with radiation therapy prior to the implementation of the MUSIC-CARE device.

DETAILED DESCRIPTION:
The retrospective phase (historical comparator) includes all patients with an initial HADS score > 7 who were treated with radiotherapy during 6 months preceding the start of the prospective study. The prospective phase involves all patients with an initial HADS score > 7 who will be treated with radiotherapy and who will benefit from music sessions (MUSIC-CARE). The study will be conducted over a fixed period of 12 months (6 months recruitment and 6 months follow-up) from the first patient receiving music sessions. Anxiety will be assessed by HADS self-questionnaires, before radiotherapy, at the end of the first week and at the end of radiotherapy. These evaluation parameters will therefore be compared to the 6-month period prior to the start of the study (retrospective phase).

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Patients undergoing radiotherapy for curative treatment
* Patients with at least 15 sessions of radiotherapy
* Patients with an anxiety score > 7 on the total A of the HADS scale at the time of medical consultation

Exclusion Criteria:

* Minor patients
* Pregnant or breastfeeding patients
* Patients with major hearing loss
* Patients with psychotic disorders
* Patients who do not understand or read the French language
* Patients under guardianship or deprived of liberty
* Patients requiring radiotherapy with respiratory servo-control (the MUSIC-CARE cannot be used due to technical constraints)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients, all cancers combined, with an initial HADS score > 7 and initiating treatment in the radiotherapy department are concerned by this study.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2023-03-26 (Actual)

PRIMARY OUTCOMES:
The main objective of the study is to evaluate the impact of the MUSIC-CARE device on the level of anxiety perceived by patients during radiotherapy. | The analysis will take place after the last visit (usual 6-month visit) of the last included patient, i.e. 6 months after the end of treatment of the last patient, and within a maximum of one year after this visit.
  Perceived anxiety will be measured by the anxiety score (total A), assessed with the Hospital Anxiety and Depression Scale (HADS). To screen for anxiety symptomatology, the following interpretation is: Total A score at 7 or less: no symptomatology, Total A score of 8 to 10: questionable symptomatology, and Total A score equal to 11 and above: definite symptomatology. Anxiety will be assessed at the medical consultation, after 5 sessions and at the end of the treatment. The patients' score after 5 sessions will be used as the primary endpoint to evaluate the impact of the to evaluate the impact of the device.

CONTACTS AND LOCATIONS:
Overall Officials: Coralie Hulot, Principal Investigator — Centre de Lutte contre le Cancer Eugène Marquis
Locations (1):
- Centre de Lutte contre le Cancer Eugène Marquis, Rennes, Brittany Region, France

IPD SHARING:
Plan to Share IPD: No